CLINICAL TRIAL: NCT00754702
Title: Vinorelbine Metronomic Plus Lapatinib as Salvage Therapy for Patients With Overexpressing HER-2 Metastatic Breast Cancer. A Multicenter Phase II Study
Brief Title: Vinorelbine Metronomic Plus Lapatinib for Overexpressing HER-2 Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, Vassilis Georgoulias, MD, MD, University Hospital of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.27
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: Vinorelbine metronomic-lapatinib; Chemotherapy; Targeted therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Vinorelbine metronomic/Lapatinib
  Interventions: Drug: Vinorelbine; Drug: Lapatinib

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine p.o (50 mg 3 times a week) until disease progression or appearance of unacceptable toxicity
  Other Names: Navelbine
Drug: Lapatinib — Lapatinib p.o every day without interruption disease progression or appearance of unacceptable toxicity
  Other Names: Tyverb; Tykerb

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of metronomic oral vinorelbine taken three times a week plus daily lapatinib without break, as salvage treatment in patients with metastatic breast cancer.

DETAILED DESCRIPTION:
Continuous administration of oral vinorelbine, given three times a week (metronomic) is feasible and exceptionally well tolerated at doses up to 50 mg. Early results show activity against refractory tumors and provide evidence towards clinical proof of efficacy for metronomic chemotherapy. Recently, lapatinib plus capecitabine was proven superior to capecitabine alone in women with HER2-positive advanced breast cancer that has progressed after treatment with regimens that included an anthracycline, a taxane, and trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically- confirmed metastatic breast adenocarcinoma
* Age 18-75 years
* HER2 status positive according to the local institution reported grade 3+ staining intensity (on a scale of 0 to 3) by means of immunohistochemical analysis or grade 2+ staining intensity by means of immunohistochemical analysis with gene amplification on fluorescence in situ hybridization
* Previous therapies had to include, regimens containing an anthracycline and a taxane
* Previous treatment with trastuzumab, alone or in combination with chemotherapy for locally advanced or metastatic disease, is required
* Measurable disease as defined by the presence of at least one measurable lesion (except bone metastases, ascites or pleural effusions)
* Performance status (WHO) 0-2
* Adequate liver (serum bilirubin <1.5 times the upper normal limit; AST and ALT <2.5 times the upper normal limit in the absence of demonstrable liver metastases, or <5 times the upper normal limit in the presence of liver metastases); adequate renal function (serum creatinine <1.5 times the upper normal limit); and bone marrow (neutrophils ≥ 1.5x 109 /L, and platelets ≥ 100x 109 /L) function
* No radiation of measurable disease (except brain metastases)
* No progressive brain metastases according to clinical or radiological criteria
* No brain metastases without prior radiation therapy
* Written informed consent

Exclusion Criteria:

* Patient unable to take oral medication
* Active infection
* History of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* Other invasive malignancy except nonmelanoma skin cancer
* Psychiatric illness or social situation that would preclude study compliance
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 3 - 6 month

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
Toxicity profile | 21 days
Overall Survival | 1 year
Quality of life assessment | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (2):
- Greece (2):
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion, Crete
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens